CLINICAL TRIAL: NCT06083714
Title: Effect of Scapular Stabilization Exercises on Scoliosis Severity, Scapula Position and Shoulder Imbalance in Individuals With Adolescent Idiopathic Scoliosis
Brief Title: Effect of Scapular Stabilization Exercises in Individuals With Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Mustafa Sarı, Research Assistant, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants in this group will receive scapular stabilization exercises in addition to Schroth exercises specific to scoliosis.
  Interventions: Other: Scapular Stabilization Exercises; Other: Schroth Exercises
- Group 2 (Active Comparator): Participants in this group will receive Schroth exercises specific to scoliosis only.
  Interventions: Other: Schroth Exercises

INTERVENTIONS:
Other: Scapular Stabilization Exercises — Home-based scapular stabilization exercises (Inferior Glide, Low Row, Scapular Clock, Wall Push Up, Wall Slide and Squat Robbery) will be performed once or twice a day, 3 sets x 20 repetitions, 3 days a week for 8 weeks.
  Arms: Group 1
Other: Schroth Exercises — It will be implemented face to face, 3 days a week, each session lasting approximately 45 minutes and in 8-week programs.

SUMMARY:
Idiopathic scoliosis is a three-dimensional deformity of the spine that accounts for approximately 70% of all scoliosis anomalies, and adolescent idiopathic scoliosis (AIS) is the most common type. AIS not only changes the shape of the trunk, but also the relationships between body parts. Considering the close anatomical relationship between the scapula and the rib cage, AIS is associated with changes in scapular position and orientation. Scapular stabilization exercises; these are exercises that aim to restore the position and orientation of the scapula and the motor control and movement pattern of the muscles, thus providing scapula stability for better shoulder kinematics. There are studies reporting that scapular stabilization exercises should be included in the rehabilitation program of patients with scapular dyskinesia and various shoulder pathologies. However, no study has been found in the literature examining the effects of scapular stabilization exercises on changes in scapular position, shoulder imbalance and curve severity seen in scoliosis. Therefore, the aim of the study is to investigate the effect of scapular stabilization exercises applied in addition to Schroth exercises used in the treatment of individuals with AIS, on scoliosis severity, scapula position and shoulder imbalance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with adolescent idiopathic scoliosis,
* Having Cobb angle between 10°-30°,
* Those with main thoracic curvature,
* Risser stage between 0-3,
* Volunteer individuals

Exclusion Criteria:

* Individuals who have had surgery related to the spine and upper extremity,
* Using a supra-axillary trunk orthosis,
* Having any systemic or neurological disease

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Severity | Change from baseline at 8 weeks
  In determining the degree of curvature, the Cobb angle obtained from the spine x-ray taken in the antero-posterior direction and containing the entire spine will be accepted as the standard measurement method. End vertebral levels will be recorded on the antero-posterior x-ray. Lines perpendicular to the upper end plate of the upper end vertebra and the lower end plate of the lower end vertebra will be drawn and the angle formed between these lines will be recorded as the Cobb angle.

SECONDARY OUTCOMES:
Axial Trunk Rotation | Change from baseline at 8 weeks
  Individuals' trunk rotation angles will be measured with the Adam's Forward Bend Test, which is considered the most practical scoliosis evaluation method in the clinic.
Scapula Position-XRay | Change from baseline at 8 weeks
  Radiography measurements will be taken in the anterio-posterior direction by the same technician. Scapular position will be measured by drawing a vertical axis line connecting two points on the centerline of the sternal body. The vertical distance to the vertical axis line will be calculated separately at the superior border, at the midpoint of the vertebral border, and at the inferior border of the scapula.
Scapula Position-Lateral Scapula Slide Test | Change from baseline at 8 weeks
  It is a quantitative method developed by Kibler and used to define scapular symmetry by measuring the distance between the distal end of the scapula and the spinous process of the aligned vertebra in three different arm positions. Patients will be asked to stand steadily on a hard, flat surface. Measurements; It will be performed in 3 different positions: arms next to the body, hands on the waist, arms raised to the sides at shoulder level, and the thumb pointing to the ground. A difference of more than 1.5 cm between two edges will be considered asymmetric.
Scapula Position-Scapular Index | Change from baseline at 8 weeks
  It is obtained by measuring the distance from the sternal notch (SN) to the coracoid process (CP) and the horizontal distance from the posterolateral angle (PLA) of the acromion to the corresponding thoracic spine (TS) with a tape measure. As the final score; The formula [(distance between SN-CP / distance between PLA-TS) X 100] is used. A lower scapular index score indicates an increase in scapula internal rotation.
Periscapular Muscle Strength | Change from baseline at 8 weeks
  Isometric strength testing of the upper trapezius, middle trapezius, lower trapezius and serratus anterior muscles will be performed using a hand dynamometer as described by Kendall.
Shoulder Imbalance-Radiographic | Change from baseline at 8 weeks
  For radiographic evaluation of shoulder imbalance; coracoid height difference, clavicular angle, clavicle-rib intersection difference, radiographic shoulder height, T1 tilt, first rib angle and neck tilt measurements will be used.
Shoulder Imbalance-Clinical | Change from baseline at 8 weeks
  For clinical evaluation of shoulder imbalance; shoulder level angle, anterior/posterior axillary angle, scapular angle, shoulder height difference, trapezial and clavicular angle and trapezial area measurements will be used.
Quality of Life Related to Scoliosis | Change from baseline at 8 weeks
  It will be evaluated using the Japanese Scoliosis Questionnaire-27, which was developed by Doi et al. and its validity and reliability in Turkish was made by Bazancir et al. Ratings are on a 5-point Likert-type scale from 0 = "not at all" to 4 = "quite a bit", and the total score ranges from 0 to 108 points. A lower score indicates a better quality of life
Cosmetic Deformity | Change from baseline at 8 weeks
  The Walter Reed Visual Assessment Scale (WRVAS) is a scale consisting entirely of visual figures developed to help individuals with idiopathic scoliosis describe how they perceive their deformity. The WRVAS scale consists of 7 items that evaluate spinal deformity, costal protrusion, lumbar protrusion, thoracic deformity, trunk imbalance, shoulder asymmetry and scapular asymmetry, and include 5 different figures representing severity, showing different aspects of spinal deformity. The figures in each item are scored between 1 and 5 points according to the severity of deformity (1: no deformity, 5: severe deformity). The person marks the figure that suits his/her body in each item of the scale. The scale allows scoring of curve severity by focusing on the person's perception of posture.
Satisfaction Level | Change from baseline at 8 weeks
  Individuals' satisfaction levels with scapula and spine position and shoulder symmetry will be evaluated with a survey created by the researchers in the light of current literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Çankaya, Turkey (Türkiye)